CLINICAL TRIAL: NCT05350280
Title: Evaluation the Effects of Low-intensity Electrical Current on the Rate of Orthodontic Tooth Movement, and Dentoalveolar Changes During En-masse Retraction of Maxillary Anterior Teeth: A Randomized Controlled Clinical Trial)
Brief Title: Evaluation of the Effect of Electrical Stimulation on the Rate of Orthodontic Tooth Movement and the Dental Arches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-06-2022
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Class II Malocclusion
Keywords: Electrical stimulation; Low-intensity electrical current (LIEC); En-masse retraction; Pain; Discomfort
MeSH Terms: conditions — Overbite; Pain | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity electrical current (LIEC) (Experimental): A removable device containing a small electrical circuit will supply the required electric current for five hours a day until the completion the retraction of the upper anterior teeth.
  Interventions: Device: electric current
- Traditional fixed orthodontic appliance (Active Comparator): The maxillary arch will be levelled and aligned. (250-300) g force will be applied on each side using two NiTi springs attached between the mini-implants and the soldered hooks in a direction approximately parallel to the occlusal plane for conducting an en-masse retraction.
  Interventions: Device: Traditional treatment

INTERVENTIONS:
Device: electric current — Electric current will be applied in this group of patients using removable device.
  Arms: Low-intensity electrical current (LIEC)
Device: Traditional treatment — No acceleration method will be performed in this group.
  Arms: Traditional fixed orthodontic appliance

SUMMARY:
Thirty-eight patients requiring extraction of maxillary first premolars and maximum anchorage to retract the upper anterior teeth will participate in the study. They will be divided randomly into two groups: electrical group and control group. In each group, en-masse retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 250 g of force per side, Mini-implants will be used as an anchor unit.

The dental changes will be detected using dental casts and to evaluate the rate of teeth retraction.

DETAILED DESCRIPTION:
Prior to enrollment of each subject into the study, they will be examined completely to determine the orthodontic treatment plan. The operator will inform them about the aim of the study and ask them to provide a written informed consent.

Self-drilling titanium mini-implants (1.6mm diameter and 8mm length) will be used. They will be inserted between the maxillary second premolar and first molar at approximately 8-10mm above the archwires at the mucogingival junction and will be checked for primary stability (mechanical retention). Then the maxillary first premolar will be extracted. The maxillary arch will be levelled and aligned. The rectangular stainless steel archwires (0.019" × 0.025") with anterior 8mm height soldered hooks distal to the canines will be inserted.

A removable device containing a small electrical circuit will be applied to each patient to supply the required electric current.

Each patient in the electrical group will be asked to wear the device for five hours a day until the completion of the retraction of the upper anterior.

(250-300) g force will be applied on each side using two NiTi springs attached between the mini-implants and the soldered hooks in a direction approximately parallel to the occlusal plane for conducting an en-masse retraction. The force level will be measured every 2 weeks. Retraction will be stopped when a class I canine relationship will be achieved and a good incisor relationship will be obtained.

Dental casts will be used for the quantification of the anteroposterior movement of the anterior teeth and the first molars every 30 days until class I canine relationship will be achieved and a good incisor relationship will be obtained. Photographs of the upper casts will be taken with a central vertical projection on the occlusal plane and with a millimeter scale at the same level used to standardize and calibrate the conditions to match the casts when photographing them. Reference points will be used for upper casts study and the measurements will be calculated using the Image J computer program. To evaluate the movement of the anterior teeth: we will project the incisive edge on the median line and measure the distance from this point to the projected position of the medial end of the third palatine wrinkle on the median line.

To evaluate the movement of the first molars: we will project the mesial contact point of the first molar on the median line and measure the distance from this point to the to the projected position of the medial end of the third palatine wrinkle on the median line.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 15-27 years.
2. Class II Division 1 malocclusion:

   * Mild / moderate skeletal Class II (sagittal discrepancy angle ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
5. Patient had previous orthodontic treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of retraction | The calculation of the rate of retraction will be done once the retraction procedures has finished. Completion of this procedure is expected to occur within 6 months in the experimental group and 8 months in the control group.
  Assessment will be performed on study models. The amount of distance being retracted in millimeters will be divided by the duration of retraction in weeks to give an estimation of the retraction rate.
Change in Incisors' positions | T0: 1 day before the beginning of retraction. T1: after 1 month (m) of retraction. T2: after 2 m of retraction. T3: after 3 m. T4: after 4 m. T5: at the end of retraction (expected to be within 6 m in the exp. group and 8 m in the control group)
  Amount of distance being traveled by the retracted anterior teeth is going to be measured on study models taken at monthly intervals until the end of the retraction phase.

SECONDARY OUTCOMES:
Change in Molars' positions | T0: 1 day before the beginning of retraction. T1: after 1 month (m) of retraction. T2: after 2 m of retraction. T3: after 3 m. T4: after 4 m. T5: at the end of retraction (expected to be within 6 m in the exp. group and 8 m in the control group)
  Amount of distance being traveled by the first molars and is going to be measured on study models taken at monthly intervals until the end of the retraction phase.
Change in the inter-canine width | T0: 1 day before the beginning of retraction. T1: after 1 month (m) of retraction. T2: after 2 m of retraction. T3: after 3 m. T4: after 4 m. T5: at the end of retraction (expected to be within 6 m in the exp. group and 8 m in the control group)
  The change in the inter-canine width (mm/month) in each group will be calculated. Assessment will be performed on the dental casts by measuring the distance between the cusp tips of the two upper canines.
Change in the inter-molar width | T0: 1 day before the beginning of retraction. T1: after 1 month (m) of retraction. T2: after 2 m of retraction. T3: after 3 m. T4: after 4 m. T5: at the end of retraction (expected to be within 6 m in the exp. group and 8 m in the control group)
  The change in the inter-molar width (mm/month) in each group will be calculated. Assessment will be performed on the dental casts by measuring the distance between the central groove of the two first maxillary molars.

CONTACTS AND LOCATIONS:
Overall Officials: Rashad I. Shaadouh, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS MSc PhD, Study Director — Department of orthodontics, Damascus University, Syria; Ghiath Mahmoud, DDS MSc PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spadari GS, Zaniboni E, Vedovello SA, Santamaria MP, do Amaral ME, Dos Santos GM, Esquisatto MA, Mendonca FA, Santamaria M Jr. Electrical stimulation enhances tissue reorganization during orthodontic tooth movement in rats. Clin Oral Investig. 2017 Jan;21(1):111-120. doi: 10.1007/s00784-016-1759-6. Epub 2016 Feb 26. PMID 26917494
- [Background] Kalemaj Z, DebernardI CL, Buti J. Efficacy of surgical and non-surgical interventions on accelerating orthodontic tooth movement: a systematic review. Eur J Oral Implantol. 2015 Spring;8(1):9-24. PMID 25738176
- [Background] Zaniboni E, Bagne L, Camargo T, do Amaral MEC, Felonato M, de Andrade TAM, Dos Santos GMT, Caetano GF, Esquisatto MAM, Santamaria M Jr, Mendonca FAS. Do electrical current and laser therapies improve bone remodeling during an orthodontic treatment with corticotomy? Clin Oral Investig. 2019 Nov;23(11):4083-4097. doi: 10.1007/s00784-019-02845-9. Epub 2019 Feb 15. PMID 30771000
- [Background] Jing D, Xiao J, Li X, Li Y, Zhao Z. The effectiveness of vibrational stimulus to accelerate orthodontic tooth movement: a systematic review. BMC Oral Health. 2017 Dec 1;17(1):143. doi: 10.1186/s12903-017-0437-7. PMID 29195495
- [Background] Cadenas de Llano-Perula M, Yanez-Vico RM, Solano-Reina E, Palma-Fernandez JC, Iglesias-Linares A. Effectiveness of Biology-Based Methods for Inhibiting Orthodontic Tooth Movement. A Systematic Review. J Clin Pediatr Dent. 2017;41(6):494-502. doi: 10.17796/1053-4628-41.6.14. Epub 2017 Sep 22. PMID 28937886
- [Derived] Shaadouh RI, Hajeer MY, Awawdeh MA, Jaber ST, Mahmoud GA, Almasri IA. Effectiveness of low-intensity electrical current in accelerating the en-masse retraction of the upper anterior teeth following first-premolar extraction in young adult patients with Class II division 1 malocclusion: A randomized controlled clinical trial. Int Orthod. 2024 Dec;22(4):100921. doi: 10.1016/j.ortho.2024.100921. Epub 2024 Sep 23. PMID 39316889